CLINICAL TRIAL: NCT01986738
Title: A Pilot Trial to Determine the Extent of Inter- and Intra-Treatment Organ Motion Using Active Breathing Control Device (ABC) in Patients With Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2011.055; HUM00050677 (Other: University of Michigan); NCT01832142 (obsolete NCT alias)
Record Dates: First submitted 2013-10-29; First posted 2013-11-18 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Radiation Treatment: Patients undergoing standard of care radiation treatment with Active Breathing Control (ABC)
  Interventions: Radiation: Standard Radiation Therapy; Device: Active Breathing Control Device (ABC); Device: Computed Tomography Scan (CT)

INTERVENTIONS:
Radiation: Standard Radiation Therapy — Radiotherapy will be planned and delivered according to institutional standard of care.
Device: Active Breathing Control Device (ABC)
Device: Computed Tomography Scan (CT)

SUMMARY:
This is a study to assess the motion of pancreatic tumors during radiation therapy using Computed Tomography (CT) Scans and an Active Breathing Control (ABC) Device.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* A working diagnosis (with or without histologic confirmation) of pancreatic cancer
* A plan to treat with radiotherapy (or chemoradiotherapy)
* Patients must have fiducial marker(s) endoscopically placed within the pancreas for clinical treatment.

Exclusion Criteria:

* Previous abdominal radiotherapy.
* Patients with a history of major abdominal surgery.
* Patients who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pancreatic cancer patients undergoing radiation treatment with active breathing control will be asked if they would like to participate.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Distance traveled by the pancreatic tumor during radiation treatment using Computed Tomography (CT) Scans and an Active Breathing Control (ABC) Device | Weeks -3 to -1, Week 1, Week 3, Week 5
  A marker (implanted near the radiation site, prior to treatment, as a point of reference) will be noted in space on an x, y and z plane using a CT scan. The excursion of this marker during treatment will be determined and the distance traveled, as well as the overall vector (distance and magnitude), will be calculated. Later scans will assess changes in the ability to calculate distance traveled and overall vector of travel.
Distance traveled by the pancreatic tumor between radiation treatments using Computed Tomography (CT) Scans and an Active Breathing Control (ABC) Device | Week -3 to -1, Week 1, Week 3, Week 5
  A marker (implanted near the radiation site prior to treatment as a point of reference) will be noted in space on an x, y and z plane on a pre-treatment/planning Computed Tomography (CT) scan. The relative position of the marker on later CT scans will be compared to the pre-treatment/planning scan and the difference in position will be calculated. The change in the position between all CT scans will be calculated for statistical analysis of tumor movement while undergoing treatment with an Active Breathing Control (ABC) Device.

SECONDARY OUTCOMES:
Probability of surrounding normal tissue being a particular distance from the tumor marker at any time point. | Week -1 to -3, Week 1, Week 3, Week 5
Assess the impact of the determined treatment margins on the radiation dose to normal tissues and the ability to escalate dose to the tumor using Intensity-Modulated Radiation Therapy (IMRT) | Analysis will take place after treatment at approximately week 6
  To assess the impact of the determined treatment margins on radiation dose distribution, we will retrospectively recalculate the patient's treatment plan based on the measured motion of the tumor and normal tissue. This new treatment plan will be compared with the original treatment plan. If the new treatment plan suggests normal tissue was exposed to a reduced amount of radiation, multiple treatment plans will be generated to assess the extent to which this reduction will allow for increased tumor dose in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Cuneo, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States